CLINICAL TRIAL: NCT00156078
Title: A 14-Week, Double-Blind, Randomized, Placebo-Controlled, Multicenter Study To Evaluate The Safety And Efficacy Of Pregabalin (150mg-600mg/Day) Using A Flexible Optimal Dose Schedule In Patients With Painful Diabetic Peripheral Neuropathy (DPN).
Brief Title: A Study To Evaluate Pregabalin In Patients With Painful Diabetic Peripheral Neuropathy (DPN)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081030
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2008-03

CONDITIONS: Diabetic Neuropathy, Painful
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Pregabalin

INTERVENTIONS:
Drug: pregabalin

SUMMARY:
A study of pregabalin efficacy and safety in a racially and culturally diverse group of subjects with painful diabetic peripheral neuropathy (DPN).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 1 or 2 diabetes mellitus.
* Diagnosis of painful DPN for at least 12 months but less than 5 years in duration.

Exclusion Criteria:

* Neurologic Disorders unrelated to diabetic neuropathy that may confuse or confound the assessment of neuropathic pain.
* Presence of any severe pain associated with conditions other than DPN that may confuse or confound the assessment of neuropathic pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450
Dates: Start 2005-01; Study Completion 2007-05

PRIMARY OUTCOMES:
Mean pain score

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (35):
- Pfizer Investigational Site, Buenos Aires, Argentina
- Brazil (2):
  - Pfizer Investigational Site, Belo Horizonte, Minas Gerais
  - Pfizer Investigational Site, Niterói, Rio de Janeiro
- Chile (2):
  - Pfizer Investigational Site, Valparaíso, Región de Valparaíso
  - Pfizer Investigational Site, Providencia, Santiago Metropolitan
- Colombia (2):
  - Pfizer Investigational Site, Medellín, Antioquia
  - Pfizer Investigational Site, Bogotá, Cundinamarca
- Pfizer Investigational Site, Quito, Pichincha, Ecuador
- Indonesia (2):
  - Pfizer Investigational Site, Jakarta Pusat
  - Pfizer Investigational Site, Surabaya
- Pfizer Investigational Site, Amman, Jordan
- Pfizer Investigational Site, Beirut, Lebanon
- Pfizer Investigational Site, Kuala Lumpur, Malaysia
- Mexico (3):
  - Pfizer Investigational Site, Monterrey, Nuevo León
  - Pfizer Investigational Site, Mexico City
  - Pfizer Investigational Site, San Luis Potosí City
- Philippines (2):
  - Pfizer Investigational Site, España, Manila
  - Pfizer Investigational Site, Quezon City
- Pfizer Investigational Site, Riyadh, Saudi Arabia
- Pfizer Investigational Site, Singapore, Singapore
- South Korea (2):
  - Pfizer Investigational Site, Pusan
  - Pfizer Investigational Site, Seoul
- Taiwan (2):
  - Pfizer Investigational Site, Gueishan Shiang, Taoyan Hsien
  - Pfizer Investigational Site, Taipei
- Thailand (2):
  - Pfizer Investigational Site, Khet Rajathevee, Bangkok
  - Pfizer Investigational Site, Muang, Chiang Mai
- Turkey (Türkiye) (5):
  - Pfizer Investigational Site, Çapa, Istanbul
  - Pfizer Investigational Site, Ankara
  - Pfizer Investigational Site, Istanbul
  - Pfizer Investigational Site, Izmir
  - Pfizer Investigational Site, Mersin
- Pfizer Investigational Site, Abu Dhabi, United Arab Emirates
- Venezuela (2):
  - Pfizer Investigational Site, El Hatillo Municipality, Caracas-Estado Miranda
  - Pfizer Investigational Site, Caracas, Distrito Federal
- Pfizer Investigational Site

REFERENCES:
- [Derived] Alexander J Jr, Edwards RA, Manca L, Grugni R, Bonfanti G, Emir B, Whalen E, Watt S, Brodsky M, Parsons B. Integrating Machine Learning With Microsimulation to Classify Hypothetical, Novel Patients for Predicting Pregabalin Treatment Response Based on Observational and Randomized Data in Patients With Painful Diabetic Peripheral Neuropathy. Pragmat Obs Res. 2019 Oct 31;10:67-76. doi: 10.2147/POR.S214412. eCollection 2019. PMID 31802967
- [Derived] Alexander J Jr, Edwards RA, Brodsky M, Manca L, Grugni R, Savoldelli A, Bonfanti G, Emir B, Whalen E, Watt S, Parsons B. Using time series analysis approaches for improved prediction of pain outcomes in subgroups of patients with painful diabetic peripheral neuropathy. PLoS One. 2018 Dec 6;13(12):e0207120. doi: 10.1371/journal.pone.0207120. eCollection 2018. PMID 30521533
- [Derived] Edwards RA, Bonfanti G, Grugni R, Manca L, Parsons B, Alexander J. Predicting Responses to Pregabalin for Painful Diabetic Peripheral Neuropathy Based on Trajectory-Focused Patient Profiles Derived from the First 4 Weeks of Treatment. Adv Ther. 2018 Oct;35(10):1585-1597. doi: 10.1007/s12325-018-0780-3. Epub 2018 Sep 11. PMID 30206821
- [Derived] Parsons B, Li C, Emir B, Vinik AI. The efficacy of pregabalin for treating pain associated with diabetic peripheral neuropathy in subjects with type 1 or type 2 diabetes mellitus. Curr Med Res Opin. 2018 Nov;34(11):2015-2022. doi: 10.1080/03007995.2018.1509304. Epub 2018 Sep 20. PMID 30084288
- [Derived] Markman JD, Jensen TS, Semel D, Li C, Parsons B, Behar R, Sadosky AB. Effects of Pregabalin in Patients with Neuropathic Pain Previously Treated with Gabapentin: A Pooled Analysis of Parallel-Group, Randomized, Placebo-controlled Clinical Trials. Pain Pract. 2017 Jul;17(6):718-728. doi: 10.1111/papr.12516. Epub 2016 Dec 1. PMID 27611736
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081030&StudyName=A+Study+To+Evaluate+The+Safety+And+Efficacy+Of+Pregabalin+In+Patients+With+Painful+Diabetic+Peripheral+Neuropathy+%28DPN%29%2E